CLINICAL TRIAL: NCT04890600
Title: Investigation on Psycological Well-being in Healthcare Workers of San Raffaele Institution During COVID-19 Emergency Context
Brief Title: COVID-19 and Psycological Well-being in Healthcare Workers
Acronym: BE-STRONG
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 20/14
Record Dates: First submitted 2021-04-22; First posted 2021-05-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2021-05

CONDITIONS: Distress, Emotional; Coping Behavior
Keywords: COVID-19, resilience, depression, healthcare workers
MeSH Terms: conditions — COVID-19; Depression

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: well-being assessment — exploration of emotional, cognitive and behavioural resources of healthcare professionals

SUMMARY:
Well-being of healthcare workers is assessed by specific questionaries validated for resilience, depression, anxiety, coping strategies and fear for COVID-19.

After signing informed consent and privacy informed consent subject are asked to complete questionaries presented as google modules.

No personal data are required.

DETAILED DESCRIPTION:
Well-being of healthcare workers is assessed by specific questionaries validated for resilience, depression, anxiety, coping strategies and fear for COVID-19.

Data will be analysed to investigate levels of resilience in healthworkers that have been in contact with patients or relatives with COVID-19.

Intervention strategies engaged by subjects are monitored to understand unmet feedings to promote well-being.

ELIGIBILITY:
Inclusion Criteria:

* Healthworkers of San Raffaele Institution
* age>18

Exclusion Criteria:

* all those who do not agree

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: nurses, medical doctors, therapists, researchers, administrative workers
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Levels of anxiety and depression | 6 months
  Hospital Anxiety and Depression Scale (HADS) Consists of 14 questions, each of which is rated from 0 to 4 according to the severity of the experienced symptoms.
Coping strategies | 6 months
  Brief-COPE Consists of 28 items divided into 14 scales, relating to 14 identified coping strategies. Each item is rated on a 4 points Likert scale.
Levels of resilience | 6 months
  14-Item Resilience Scale Consists of 14 items, each rated on a 7 levels Likert scale and evaluates the levels of resilience.
Levels of fear of COVID-19 | 6 months
  FEAR OF COVID-19 SCALE Consists of 7 items, each rated on a Likert scale from 1 to 5, with the aim of assessing the levels of fear related to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bonassi, PhD, Principal Investigator — IRCCS San Raffaele Roma
Locations (1):
- IRCCS San Raffaele Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No